CLINICAL TRIAL: NCT01563315
Title: Community-acquired Pneumonia: A Prospective Observational Study to Explore Etiology, Risk Factors and Potential Predictors for re- Admittance to Hospital and All-cause Mortality
Brief Title: Community-acquired Pneumonia in Buskerud County in Norway
Status: Completed | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Vestre Viken HF - Buskerud Hospital (Unknown); Oslo University Hospital (Other); UMass Medical school, Massachusetts - USA (Unknown)
Responsible Party: Sponsor
Other Study IDs: REK:S-06266a
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Community-Acquired Infections; Pneumonia
Keywords: Community-Acquired Infections; Pneumonia/microbiology; Pneumonia/diagnosis; Prognosis; Prospective Studies
MeSH Terms: conditions — Community-Acquired Infections; Pneumonia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, blood culture, airways specimens, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adults with CAP admitted to hospital: All adult patients with CAP admitted to Vestre Viken HF-Buskerud Hospital (VVHF-BH), a 400-bed community general hospital, between January 2008 og January 2011 were evaluated for inclusion in the study.

SUMMARY:
The purpose of this study is to determine the etiology of community-acquired pneumonia, to assess risk factors and to investigate potential prognostic biomarkers of serious disease and fatal outcome.

DETAILED DESCRIPTION:
Background: This project addresses an important challenge in international medicine: Pneumonia as the leading cause of death from infection in developed countries. Purpose: (A) Determine the etiology of CAP among adult hospitalized patients- especially the occurrence of mixed infections- by systematic implementation of combined conventional and new diagnostic methods. (B) Assess risk factors of CAP, such as COPD, congestive heart failure, smoking, malignancy etc., predictive of re-admittance to hospital and mortality. (C) Examine the prognostic value of potential predictors in relation to all-cause mortality in adult patients hospitalized with CAP. Design: Prospective observational study with inclusion of 270 adult patients during a 3-year period, who all required admission for pneumonia in a community hospital setting. Clinical and biochemical data was recorded longitudinally by inclusion, at stable clinical situation and after 6 weeks, and mortality and need for re-admission within 12 months. Patients were examined systematically, using modern research methods to explore relevant microbes. At all points, blood tests were sampled for clinical-chemical analysis, DNA, RNA and immunological analyses. Application: A translational research approach with the ambitions to elucidate new pathogenic mechanisms which could lead to new diagnostic tools and treatment modalities. This will possibly lead to less drug exposure and unnecessary hospitalization both of which have positive consequences for patients and medical care costs.

ELIGIBILITY:
Inclusion Criteria:

* New infiltrate on chest X-ray and
* Fever > 38,0 by rectal measurement

  * at least one of these additional criteria: Cough +/- expectoration, dyspnoea, respiratory chest pain, crackles or reduced respiratory sounds.
* Criteria must be present within 48 hours after admission

Exclusion Criteria:

* Patients < 18 years
* Non infectious cause of lung infiltration (tumors, embolism)
* Bronchial obstruction (tumor, bronchiectasia)
* Hospitalised more than 48 hours or discharged within the last 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with CAP admittet to Vestre Viken HF-Buskerud Hospital (VVHF-BH) between January 2008 og January 2011, were evaluated for inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
all cause mortality | one year

SECONDARY OUTCOMES:
Re-admission to hospital | One month

CONTACTS AND LOCATIONS:
Overall Officials: Lars Heggelund, MD, PhD, Study Director — Vestre Viken Hospital Trust and Oslo University Hospital; Einar Husebye, MD, PhD, Study Chair — Vestre Viken Hospital Trust; Jan C Holter, MD, Principal Investigator — Vestre Viken Hospital Trust
Locations (1):
- Vestre Viken Hospital Trust, Drammen, Buskerud, Norway

REFERENCES:
- [Derived] Holter JC, Muller F, Bjorang O, Samdal HH, Marthinsen JB, Jenum PA, Ueland T, Froland SS, Aukrust P, Husebye E, Heggelund L. Etiology of community-acquired pneumonia and diagnostic yields of microbiological methods: a 3-year prospective study in Norway. BMC Infect Dis. 2015 Feb 15;15:64. doi: 10.1186/s12879-015-0803-5. PMID 25887603